CLINICAL TRIAL: NCT07106177
Title: Three-dimensional Accuracy of Direct Digital Scanning for All on Four Implants in Comparison to a Custom-made Verification Jig in Fully Edentulous Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yasser Ahmed (Other)
Collaborators: Alexandria University (Other)
Responsible Party: Sponsor-Investigator, Yasser Ahmed, Associate Professor of Fixed Prosthodontics, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1093-05/2025
Record Dates: First submitted 2025-07-22; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Edentulism

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Scanning with the aid of jig (Experimental)
  Interventions: Other: Scanning with verification jig
- Scanning without jig (Active Comparator)
  Interventions: Other: Direct intraoral scanning

INTERVENTIONS:
Other: Scanning with verification jig — Comparing Relative Implant Positions of the 4 implants in each case obtained through desktop scanning of intraoral provisional verification jig. All-on-4 treatment for mandibular and maxillary edentulous cases were scanned using the Medit i700 intraoral scanner. Scan data were imported into Exocad software, where scan-body matching was performed using the Neodent library to determine the positions of multiunit abutment analogues.
  Arms: Scanning with the aid of jig
Other: Direct intraoral scanning — Comparing Relative Implant Positions of the 4 implants in each case obtained through direct intraoral scanning without jig. All-on-4 treatment for mandibular and maxillary edentulous cases were scanned using the Medit i700 intraoral scanner. Scan data were imported into Exocad software, where scan-body matching was performed using the Neodent library to determine the positions of multiunit abutment analogues.
  Arms: Scanning without jig

SUMMARY:
The aim of this study is to assess the three-dimensional accuracy of direct intraoral scanning in All-on-4 implant-supported prostheses by comparing intraoral scan data with a custom-made verification jig.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complete mandibular edentulism.
* Patients requiring full-arch rehabilitation with an All-on-4 implant concept.
* Absence of systemic conditions that could affect bone healing or osseointegration.
* Adequate bone volume in the anterior mandible for implant placement without the need for additional grafting.
* Patients capable of maintaining oral hygiene

Exclusion Criteria:

* Patients with uncontrolled systemic diseases (e.g., diabetes, osteoporosis).
* History of head and neck radiation therapy.
* Severe parafunctional habits (e.g., bruxism).
* Patients with inadequate bone volume requiring extensive grafting procedures.
* Active periodontal or oral infections.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-07-10 (Actual); Study Completion 2025-07-10 (Actual)

PRIMARY OUTCOMES:
Vertical Deviation | through study completion, an average of 1 year
  Analogues Saved from the Intraoral scan and those saved from stone model were superimposed. The vertical discrepancy (mm) in implant position between intraoral digital scanning and verification jig-based stone model in All-on-4 implant cases.
Angular deviation | through study completion, an average of 1 year
  Analogues Saved from the Intraoral scan and those saved from stone model were superimposed. The angular difference (degrees) in implant position between intraoral digital scanning and verification jig-based stone model in All-on-4 implant cases.
Horizontal deviation | through study completion, an average of 1 year
  Analogues Saved from the Intraoral scan and those saved from stone model were superimposed. The horizontal discrepancy (mm) in implant position between intraoral digital scanning and verification jig-based stone model in All-on-4 implant cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt